CLINICAL TRIAL: NCT06953076
Title: MyomaS Aspect Transformation at Ultrasound During Relugolix Estradiol Noretisterone Treatment: MySaturn Study
Brief Title: Ultrasound Transformation of Myomas During Relugolix-Estradiol-Norethisterone Treatment: The MySaturn Study
Acronym: MySaturn
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, ROMUALDI DANIELA, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7427
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Uterine Bleeding; Uterine Leiomyomas; Uterine Hemorrhage; Uterine Neoplasms
Keywords: myomas; uterine bleeding; fibroids; relugolix; ormonal therapy; smooth muscle cells tumor
MeSH Terms: conditions — Uterine Hemorrhage; Myofibroma; Uterine Neoplasms; Myoma; Leiomyoma | interventions — relugolix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Uterine fibroids symptomatic for abnormal uterine bleeding: Patients with ultrasound diagnosis of uterine fibroids, symptomatic for abnormal uterine bleeding, eligible for oral medical therapy with relugolix/estradiol/norethisterone
  Interventions: Drug: Relugolix/estradiol/norethisterone acetate

INTERVENTIONS:
Drug: Relugolix/estradiol/norethisterone acetate — Oral therapy administered to patients with symptomatic uterine fibroids presenting with abnormal uterine bleeding
  Other Names: Ryeqo

SUMMARY:
Uterine fibroids are benign tumors originating from the uterine muscle, affecting up to 70% of women by their 50s. Risk factors include African descent, nulliparity, obesity, and diabetes. While many fibroids are asymptomatic, 25-50% of affected women experience symptoms like heavy menstrual bleeding, pelvic pain, and pressure-related issues. Accurate diagnosis and differentiation from rare malignant tumors (e.g., uterine sarcomas) remain challenging, particularly before surgery.

Ultrasound is the first-line tool for evaluating fibroids, with specific features (e.g., shape, vascularity) helping distinguish benign from suspicious lesions. The MUSA guidelines standardize ultrasound terminology for myometrial assessments. Current treatment options vary based on symptoms and malignancy risk. Among pharmacologic options, the combination of relugolix, estradiol, and norethisterone has shown efficacy in reducing bleeding and pain in symptomatic fibroids, with a favorable safety profile. However, its impact on fibroid morphology and ultrasound appearance is not yet well understood.

DETAILED DESCRIPTION:
Uterine fibroids are the most common benign tumors in women of reproductive age, affecting up to 70% of women in their 40s and 50s. While often asymptomatic, around 25-50% experience symptoms such as heavy menstrual bleeding, pelvic pain, and pressure-related issues. The severity depends on the number, size, and location of the fibroids.

Though most fibroids are benign, a small risk exists for malignant uterine tumors (e.g., leiomyosarcomas, STUMPs). Diagnosing these malignancies preoperatively remains a challenge due to the lack of reliable imaging markers. Ultrasound is the first-line diagnostic tool, guided by MUSA criteria, but further prospective data are needed to improve risk stratification.

The combination of Relugolix, Estradiol, and Norethisterone (Ryeqo®) is an effective medical treatment for symptomatic fibroids, especially in premenopausal women. It reduces bleeding while minimizing side effects of estrogen deprivation. Over 70% of women in clinical trials have shown significant improvement within 24 weeks. However, its effect on fibroid morphology and ultrasound features remains unclear.

The MySaturn Study aims to assess whether this therapy modifies the ultrasound appearance of myometrial lesions over 12 months. The study also tracks symptom changes and adverse events. It involves 111 premenopausal women in a monocentric ambispective observational design, combining retrospective and prospective data from July 1, 2023. The study spans 3 years (2 years of enrollment + 1 year follow-up) and uses routine clinical, laboratory, and imaging data for analysis.

Adverse events will be monitored and reported in accordance with national pharmacovigilance regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Pre-menopausal status.
3. Ultrasound diagnosis of benign myometrial lesion.
4. Symptomatic patients presenting with abnormal uterine bleeding (menorrhagia/metrorrhagia).
5. Availability of ultrasound images in digital format.

Exclusion Criteria:

1. Patient refusal.
2. Age < 18 years.
3. Postmenopausal women.
4. Myometrial lesion ≤ 10 mm.
5. Myometrial formation suspected of malignancy on ultrasound (e.g., STUMP - Uterine Leiomyosarcoma).
6. Asymptomatic patients with uterine fibromatosis.
7. Personal history of malignant or premalignant uterine neoplasia (e.g., STUMPs, leiomyosarcoma, atypical endometrial hyperplasia, endometrial carcinoma, cervical carcinoma).
8. Patients with ovarian pathology.
9. Patients currently undergoing treatment for another malignancy.
10. Patients lacking available digital ultrasound images or whose image quality is insufficient to adequately characterize the target lesion's ultrasound features

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with ultrasound diagnosis of uterine fibroids, symptomatic for abnormal uterine bleeding, eligible for oral medical therapy with relugolix/estradiol/norethisterone
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
To observe modifications in the volume of the myometrial lesion during treatment with relugolix/estradiol/norethisterone | at baseline, and after 3 months, 6 months, and 12 months from treatment initiation
  Modifications in the volume of the myometrial lesion
To observe the ultrasound features of myometrial lesions during treatment with relugolix/estradiol/norethisterone | at baseline, and after 3 months, 6 months, and 12 months from treatment initiation
  * Uterine volume
  * Outer contour: regular or irregular;
  * Echogenicity of the myometrial formation: mixed or homogeneous;
  * Presence of cystic areas;
  * Presence of acoustic shadows;
  * Vascularization of the lesions, expressed on a 1 to 4 ordinal scale;
  * "Cooked aspect" , if present

SECONDARY OUTCOMES:
Description of the clinical characteristics of the study population during treatment with relugolix/estradiol/norethisterone. | at baseline, and after 3 months, 6 months, and 12 months from treatment initiation
  * Effect on abnormal uterine bleeding, measured as the number of sanitary pads used during the cycle in patients who do not develop amenorrhea;
  * Hemoglobin, serum iron, and ferritin levels
  * Dyspareunia, assessed using NRS or VAS scales;
  * Chronic pelvic pain, assessed using NRS or VAS scales;
  * Compression-related symptoms;
  * Pollakiuria and dyschezia;
  * Dyspareunia

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Romualdi, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC GINECOLOGIA ONCOLOGICA, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Education and Practical Standards Committee, European Federation of Societies for Ultrasound in Medicine and Biology. Minimum training recommendations for the practice of medical ultrasound. Ultraschall Med. 2006 Feb;27(1):79-105. doi: 10.1055/s-2006-933605. No abstract available. PMID 16508866
- [Result] Al-Hendy A, Lukes AS, Poindexter AN 3rd, Venturella R, Villarroel C, Critchley HOD, Li Y, McKain L, Arjona Ferreira JC, Langenberg AGM, Wagman RB, Stewart EA. Treatment of Uterine Fibroid Symptoms with Relugolix Combination Therapy. N Engl J Med. 2021 Feb 18;384(7):630-642. doi: 10.1056/NEJMoa2008283. PMID 33596357
- [Result] Al-Hendy A, Venturella R, Arjona Ferreira JC, Li Y, Soulban G, Wagman RB, Lukes AS. LIBERTY randomized withdrawal study: relugolix combination therapy for heavy menstrual bleeding associated with uterine fibroids. Am J Obstet Gynecol. 2023 Dec;229(6):662.e1-662.e25. doi: 10.1016/j.ajog.2023.08.030. Epub 2023 Sep 2. PMID 37666383
- [Result] Al-Hendy A, Lukes AS, Poindexter AN 3rd, Venturella R, Villarroel C, McKain L, Li Y, Wagman RB, Stewart EA. Long-term Relugolix Combination Therapy for Symptomatic Uterine Leiomyomas. Obstet Gynecol. 2022 Dec 1;140(6):920-930. doi: 10.1097/AOG.0000000000004988. Epub 2022 Nov 2. PMID 36357960
- [Result] De La Cruz MS, Buchanan EM. Uterine Fibroids: Diagnosis and Treatment. Am Fam Physician. 2017 Jan 15;95(2):100-107. PMID 28084714
- [Result] Van den Bosch T, Dueholm M, Leone FP, Valentin L, Rasmussen CK, Votino A, Van Schoubroeck D, Landolfo C, Installe AJ, Guerriero S, Exacoustos C, Gordts S, Benacerraf B, D'Hooghe T, De Moor B, Brolmann H, Goldstein S, Epstein E, Bourne T, Timmerman D. Terms, definitions and measurements to describe sonographic features of myometrium and uterine masses: a consensus opinion from the Morphological Uterus Sonographic Assessment (MUSA) group. Ultrasound Obstet Gynecol. 2015 Sep;46(3):284-98. doi: 10.1002/uog.14806. Epub 2015 Aug 10. PMID 25652685
- [Result] Ciccarone F, Biscione A, Robba E, Pasciuto T, Giannarelli D, Gui B, Manfredi R, Ferrandina G, Romualdi D, Moro F, Zannoni GF, Lorusso D, Scambia G, Testa AC. A clinical ultrasound algorithm to identify uterine sarcoma and smooth muscle tumors of uncertain malignant potential in patients with myometrial lesions: the MYometrial Lesion UltrasouNd And mRi study. Am J Obstet Gynecol. 2025 Jan;232(1):108.e1-108.e22. doi: 10.1016/j.ajog.2024.07.027. Epub 2024 Jul 30. PMID 39084498
- [Result] Stewart EA, et al. Uterine fibroids. Lancet. 2022; 400(10352):1341-1351

DOCUMENTS (1):
  • Study Protocol (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT06953076/Prot_000.pdf